CLINICAL TRIAL: NCT01683019
Title: A MULTICENTER, RANDOMIZED, BLINDED, SHAM CONTROLLED, PARALLEL GROUP TRIAL TO TEST CLINICAL EFFICACY OF LOW FREQUENCY AC MAGNETIC FIELD INDUCED EEG SYNCHRONIZATION IN MAJOR DEPRESSION
Brief Title: Feasibility Study to Test Clinical Efficacy of Low Energy AC Magnetic Field to Treat Major Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wave Neuroscience (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NST#002
Record Dates: First submitted 2012-09-04; First posted 2012-09-11 (Estimated); Results first posted 2014-05-05 (Estimated); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: Major Depressive Disorder (MDD)
Keywords: Depression; magnetic field; alpha frequency; EEG; NeoSync EEG Synchronization Therapy
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes

ARMS (3):
- Active Fixed Alpha Frequency Magnetic Stimulation (Active Comparator): Sinusoidal magnetic field set to the subject's intrinsic alpha frequency (IAF).
  Interventions: Device: NeoSync EEG Synchronization Therapy
- Active Random Frequency Magnetic Stimulation (Active Comparator): Magnetic field hops to random frequencies in the alpha band (8-13Hz), once per second.
  Interventions: Device: NeoSync EEG Synchronization Therapy
- Inactive Sham Treatment (Sham Comparator): Generate sound similar to active treatment, except that no magnetic field is generated.
  Interventions: Device: Sham NeoSync EEG Synchronization Therapy

INTERVENTIONS:
Device: NeoSync EEG Synchronization Therapy — Generate low-energy sinusoidal magnetic field above the scalp with frequency equal to the subject's intrinsic alpha frequency (IAF). Treatment is 30 minutes, administered 5 days per week for 4 weeks.
  Arms: Active Fixed Alpha Frequency Magnetic Stimulation; Active Random Frequency Magnetic Stimulation
Device: Sham NeoSync EEG Synchronization Therapy — A device that looks and sounds similar to the active treatment, but no magnetic field is generated.
  Arms: Inactive Sham Treatment

SUMMARY:
This feasibility study investigates effects of EEG-based low frequency, low emission magnetic cortical stimulation in comparison to a sham treatment in subjects with moderate to severe depressive disorder.

DETAILED DESCRIPTION:
Major Depressive Disorder (MDD) is associated with functional impairment and disability, and results in a significant burden on the affected individual, his or her family, and society in general. Psychopharmacological therapy has been shown to be effective, but may be accompanied by significant side effects. The investigators propose an alternative model, based on the relationship between symptoms, brain metabolism, and neural activity as recorded with electroencephalography (EEG). Subjects with MDD often have decreased brain metabolism, accompanied by increased EEG activity in the alpha band. The investigators hypothesis is that a gentle, non-significant risk, sinusoidal magnetic field above the subject's scalp, which oscillates at precisely his or her Intrinsic Alpha Frequency (IAF) can take advantage of this relationship to reduce symptoms without the significant side effects associated with pharmaceuticals. The investigators propose a 4-week, sham controlled, randomized, double-blind multi-center feasibility study to determine the efficacy of synchronized low energy magnetic fields delivered at the subject's IAF to treat MDD. Treatment will be given concomitant to the subject's existing medication, and will occur 5 days per week at the clinical site. Target enrollment is 45 adult subjects diagnosed with MDD.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Diagnosis of MDD with HAMD-17 greater than or equal to 17
* On a stable dose of existing medication or no medication for 1 month or longer prior to the study

Exclusion Criteria:

* Diagnosed with another primary Axis I illness
* Recent history of or current substance abuse
* Clinically significant medical illness, including any thyroid disorders
* Known pregnancy and/or lactation, or intent to become pregnant during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2008-06; Primary Completion 2008-11 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Amen Clinic, Newport Beach, California, United States
- Institute of Mental Health, Peking University, Beijing, China

REFERENCES:
- [Derived] Jin Y, Phillips B. A pilot study of the use of EEG-based synchronized Transcranial Magnetic Stimulation (sTMS) for treatment of Major Depression. BMC Psychiatry. 2014 Jan 18;14:13. doi: 10.1186/1471-244X-14-13. PMID 24438321

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited at two separate psychiatric clinics. The recruitment period was between June 9, 2008 and November 5, 2008. Recruitment was accomplished through selection from the normal patient flow at the clinics.
Pre-assignment Details: Following enrollment and completion of informed consent, subjects were randomized to a treatment arm. Subjects were instructed to continue any concomitant medication throughout the treatment period. There was no wash out or transition required.
Groups:
- Active Fixed Alpha Frequency Magnetic Stimulation: Sinusoidal magnetic field set to the subject's intrinsic alpha frequency (IAF).
  NeoSync EEG Synchronization Therapy : Generate low-energy sinusoidal magnetic field above the scalp with frequency equal to the subject's intrinsic alpha frequency (IAF). Treatment is 30 minutes, administered 5 days per week for 4 weeks.
- Active Random Frequency Magnetic Stimulation: Magnetic field hops to random frequencies in the alpha band (8-13Hz), once per second.
  NeoSync EEG Synchronization Therapy : Generate low-energy sinusoidal magnetic field above the scalp with frequency equal to the subject's intrinsic alpha frequency (IAF). Treatment is 30 minutes, administered 5 days per week for 4 weeks.
- Inactive Sham Treatment: Generate sound similar to active treatment, except that no magnetic field is generated.
  Sham NeoSync EEG Synchronization Therapy : A device that looks and sounds similar to the active treatment, but no magnetic field is generated.
Period: Overall Study
Arm/Group | Active Fixed Alpha Frequency Magnetic Stimulation | Active Random Frequency Magnetic Stimulation | Inactive Sham Treatment
Started | 18 | 15 | 19
Completed | 16 | 14 | 15
Not Completed | 2 | 1 | 4
Not completed — Withdrawal by Subject | 2 | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Fixed Alpha Frequency Magnetic Stimulation | Active Random Frequency Magnetic Stimulation | Inactive Sham Treatment | Total
Number analyzed (Participants) | 18 | 15 | 19 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 0 | 1
  Between 18 and 65 years | 17 | 14 | 19 | 50
  >=65 years | 1 | 0 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.2 (15.1) | 40.7 (15.9) | 46.3 (12.7) | 43.5 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 9 | 27
  Male | 9 | 6 | 10 | 25
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 5 | 15
  China | 13 | 10 | 14 | 37

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Hamilton Depression Rating Scale (HAMD-17) at Baseline and the End of Week 4 of Treatment.
Description: Outcome measured using the Hamilton Depression Rating Scale (HAMD-17) and calculated as percent change in severity score from baseline until the end of the 4th week of treatment.
  The HAMD-17 scale ranges between 0-54, with higher numbers indicating more severe symptoms. 0-7 is generally accepted to be within the normal range (or in clinical remission), while a score of 20 or higher indicates moderate to severe depression.
Time Frame: Assessed at baseline and the end of Week 4 of treatment.
Population: 52 subjects were randomized into the study. Of those, 7 dropped in the first week due to difficulties driving to the study site. An intent-to-treat analysis was performed on the remaining 45 subjects.
Measure: Mean (Standard Error); unit: % change in HAM-D score
Arm/Group | Active Fixed Alpha Frequency Magnetic Stimulation | Active Random Frequency Magnetic Stimulation | Inactive Sham Treatment
Number analyzed (Participants) | 16 | 14 | 15
% change in HAM-D score | -53.8 (27.8) | -53.1 (26.9) | -24.2 (24.2)

ADVERSE EVENTS:
Arm/Group | Active Fixed Alpha Frequency Magnetic Stimulation | Active Random Frequency Magnetic Stimulation | Inactive Sham Treatment
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/14 | 0/15
Other Adverse Events (participants affected / at risk) | 0/16 | 0/14 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No